CLINICAL TRIAL: NCT00869219
Title: Phase 4 Study of Topical NSAID for Ophthalmologic Use: Pain Measurement After First Drop.
Brief Title: Comparison of Pain Sensation During Single Use of Two Topical Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Santa Casa de Misericordia de Santos (Other)
Responsible Party: Gustavo Teixeira Grottone, Santa Casa de Misericordia de Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCMisericordiaSantos
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Pain
Keywords: Pain; Pain after eyedrops
MeSH Terms: conditions — Pain | interventions — nepafenac; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nevanac (Active Comparator)
  Interventions: Drug: Nevanac
- Acular LS (Active Comparator)
  Interventions: Drug: Acular LS

INTERVENTIONS:
Drug: Nevanac — 1 drop of NEVANAC at random eye
  Arms: Nevanac
Drug: Acular LS — One drop of Acular LS
  Arms: Acular LS

SUMMARY:
Different case reports are showing that depending on the drug used for eye drops, it might provoke a painful sensation. Actually two leading NSAIDs are used in ophthalmology. This study is intended to provide information about this parameter concerning these two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 21 years old
* No ocular surface pathology
* Eligible for cataract surgery

Exclusion Criteria:

* Any other eye pathology other than cataract

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Pain after instilation | 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo T Grottone, MD, MBA,MSc, Principal Investigator — SCMS; João C Grottone, MD, MBA, Study Chair — SCMS
Locations (1):
- Santa Casa de Misericordia de Santos, Santos, São Paulo, Brazil